CLINICAL TRIAL: NCT04554680
Title: Phase II Clinical Trial in Radioactive Iodine-Refractory Advanced Thyroid Carcinoma Evaluating BRAF & MEK Blockade Therapy for Re-differentiation- Applying a Novel Time-Dependent Concept
Brief Title: Clinical Trial in RAI-Refractory Thyroid Carcinoma Evaluating BRAF & MEK Blockade for Re-differentiation Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TY01/04/20; 2020/00309 (Other: NHG DSRB Reference)
Record Dates: First submitted 2020-08-29; First posted 2020-09-18 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2020-08

CONDITIONS: Thyroid Cancer
Keywords: Thyroid carcinoma; re-differentiation; radioactive iodine - refractory
MeSH Terms: conditions — Thyroid Neoplasms | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Patients with progressive, metastatic or locally advanced, unresectable radioiodine (RAI)-refractory thyroid cancer of follicular cell origin with mutation involving MAPK signalling pathway, including BRAFV600E mutation or RAS mutation.
  Interventions: Drug: dabrafenib and trametinib

INTERVENTIONS:
Drug: dabrafenib and trametinib — Participants will receive systemic therapy in the form of oral tablet dabrafenib 150mg twice a day & oral tablet trametinib 2mg once a day for 1 or 4 weeks.
  Pre- & post-systemic therapy assessment of tumor iodine absorption is done using I-124 PET CT scan. Participants are prepared for this scan with intramuscular injection of thyrogen 0.9mg on 2 consequent days, followed by I-124 PET-CT scan over the next 3 days for tumoral lesional dosimetry.
  Participants are then started on systemic therapy for 1 week, followed by I-124 PET-CT scan. If at least one tumor site can attain adequate dosimetry, RAI (I-131) treatment under thyrogen stimulation will be considered. Systemic therapy will be stopped 3 days after I-131.
  If after 1 week of systemic therapy, tumors do not reach dosimetry criteria, participants will be continued on systemic therapy for a total of 4 weeks duration, followed by I-124 PET-CT scan. If tumor can attain adequate dosimetry, I-131 treatment will be considered.

SUMMARY:
Progressive and metastatic thyroid cancer patients, who no longer respond to radioactive iodine (RAI), are currently treated with long term tyrosine kinase inhibitors to control tumor growth. The investigators will study the effect of short term oral anti-cancer drug combination, called dabrafenib (BRAF inhibitor) and trametinib (MEK inhibitor), in improving thyroid cancer RAI absorption that can potentially lead to tumor shrinkage response. To assess for suitability, participant's thyroid cancer tissue taken at the time of surgery will be tested for DNA changes, such as BRAFV600E, RAS, or MEK mutations.

Based on experimental studies, the response to these medications could occur within 1 week of treatment. So in the study, the investigators will find out whether participant's cancer would respond to 1 week of treatment with these medications rather than the 1 month duration of treatment in previous re-differentiation clinical trials. After 1 week of treatment with dabrafenib and trametinib, iodine absorption I-124 PET-CT scan will predict if the cancer will respond to RAI. If iodine absorption is insufficient on the scan, treatment with dabrafenib and trametinib will be continued for a total of 4 weeks. Then iodine absorption response of participant's cancer will be assessed on I-124 PET-CT scan again. If the iodine absorption is good at 1 week or 4 weeks, the investigators will treat the participant with thyroid cancer using RAI.

The 1-week treatment regime can potentially save cost, avoid drug toxicity with prolonged treatment, and prevent drug resistance that can occur with longer treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be at least 21 years of age on the day of signing informed consent.
2. The participant (or legally acceptable representative if applicable) provides written consent for the trial.
3. Eastern Cooperative Oncology Group (ECOG) performance status < 2
4. . The histology of the thyroid carcinoma for inclusion includes any of the following:

   * Papillary thyroid carcinoma
   * Follicular thyroid carcinoma
   * Hurthle cell carcinoma
   * Poorly differentiated thyroid carcinoma
5. Patients with a thyroid carcinoma of follicular cell origin with mutation involving MAPK signalling pathway, including BRAFV600E mutation or RAS mutation detected in a Clinical Laboratory Improvement Amendments (CLIA)-certified or US Food and Drug Administration-approved assay.
6. The patients need to fulfil one of the following criteria for RAI-refractory disease (Tuttle et al, 2019;):

   1. No 131-I uptake is present on a diagnostic 131-I scan
   2. No 131-I uptake is present on a 131I scan performed several days after 131-I therapy
   3. 131-I uptake is only present in some but not other tumor foci
   4. DTC metastasis(es) progress despite 131-I uptake
   5. DTC metastasis(es) progress despite a cumulative 131-I activity of >600 mCi
7. The metastatic tumoral lesion should have no RAI uptake on therapeutic or diagnostic radioiodine scan performed before enrolment. Alternatively, the RAI-avid metastatic lesion should not show size reduction (either remained stable in size or progressed) despite RAI therapy >6 months before study entry.
8. The disease should be measurable based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
9. Adequate haematological, renal and liver function defined as:

   1. Absolute neutrophil count (ANC) ≥ 1.5 ×109/L.
   2. Hemoglobin ≥ 9.0 g/dl (Note: The use of transfusion or other intervention to achieve hemoglobin ≥ 9.0 g/dl is acceptable).
   3. Platelets ≥ 75 ×109/L.
   4. Total bilirubin ≤2.5 x institutional upper limit of normal (unless due to Gilbert's disease).
   5. Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) / alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 x institutional upper limit of normal.
   6. Serum creatinine ≤ 1.5 x institutional upper limit of normal.
   7. Prothrombin time (PT) within the normal range for the institution.
10. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP) OR
    2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 4 months after the last dose of dabrafenib and trametinib. Contraception has to be continued for 6 months after radioactive iodine if this were to be administered. Barrier method of contraception is preferred as dabrafenib may decrease serum estrogen and progestin concentrations.

    Female patients of childbearing potential are required to have a negative serum pregnancy test within 14 days prior to the first dose of study medication.
11. A male participant must agree to use a contraception during the treatment period and for at least 4 months days after the last dose of dabrafenib and trametinib (and radioactive iodine if administered), and refrain from donating sperm during this period.

Exclusion Criteria:

Patients will not be recruited if they meet the following criteria:

1. Anaplastic thyroid carcinoma
2. Exceeded cumulative I-131 treatment dose of >600mCi
3. Treatment with I-131 therapy 6 months before study treatment.
4. G6PD deficiency due to risk of haemolytic anaemia with dabrafenib
5. Had received prior systemic anti-cancer therapy, including investigational agents within 2 weeks prior to randomisation.
6. Had received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities.
7. Patients who have not recovered from adverse events related to prior therapy for cancer to Common Terminology Criteria for Adverse Events (CTCAE) 4.03 grade 2 or less, except for alopecia.
8. Patients with a history of other active malignancy requiring cancer treatment.
9. Patients with uncontrolled brain metastases. Patients who are on a stable dose of corticosteroids for more than 1 week or off corticosteroids for 2 weeks prior to study enrolment can be enrolled.
10. On concurrent prohibitive drugs such as enzyme-inducing anti-epileptic drugs. [Refer to section 3.7 (concomitant treatment) for list of medications that require closer monitoring.]
11. Patients with a known history of retinal vein occlusion, central serous retinopathy, uncontrolled glaucoma or ocular hypertension.
12. Patients with class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
13. Corrected QT (QTc) interval greater than or equal to 480 msecs (>= 500 msec for subjects with Bundle Branch Block).
14. Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring intravenous antibiotics, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
15. Pregnant women and nursing women are excluded from this study because dabrafenib has the potential for teratogenic or abortifacient effects. In embro-fetal developmental studies in rats, developmental toxicities including reduced fetal body weight, embryo-lethality, cardiac ventricular septal defect malformations, delayed skeletal development and variation in thymic shape have been observed.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-12-30 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants attaining at least one tumor lesion with lesional dosimetry of >=2000 cGy with I-131 dose of =<300 mCi. | 1 month after start of dabrafenib and trametinib
  The primary endpoint can be considered attained in both groups of participants:
  * those that attain target lesional dosimetry after 1 week of therapy
  * those that attain target lesional dosimetry after 4 weeks of therapy

SECONDARY OUTCOMES:
Progression-free survival and overall survival | From the start of assessment until study completion, an average of 2 years
Best tumor response as assessed by RECIST criteria | From the start of assessment until study completion, an average of 2 years
Change in serum thyroglobulin level after radioactive iodine (RAI) treatment compared to baseline, pre-treatment level | 6 months after RAI treatment
The proportion of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From the start of assessment until study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore